CLINICAL TRIAL: NCT00883792
Title: NordICC The Northern-European Initiative on Colorectal Cancer
Brief Title: The Northern-European Initiative on Colorectal Cancer
Acronym: NordICC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Maria Sklodowska-Curie National Research Institute of Oncology (Other); Erasmus Medical Center (Other); Landspitali University Hospital (Other); Uppsala University Hospital (Other); Karolinska Institutet (Other); Memorial Sloan Kettering Cancer Center (Other); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Michael Bretthauer, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NordICC
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Colonoscopy screening (Experimental): One-time colonoscopy is the screening tool used in this trial. All individuals in the screening group will be offered a full colonoscopy. At colonoscopy, all detected CRC precursor lesions will be removed, whenever possible.
  Interventions: Procedure: Colonoscopy
- Control (No Intervention): The control group will not be offered any screening or intervention within the trial, but follow usual care in the participating countries. Individuals assigned to the control group will not be informed about their status as controls in the trial. This approach facilitates a truly population-based study, which will be used to estimate the effect of the screening intervention in the general population, mimicking national CRC screening programs.
  All ethics committees at the participating centres have approved the study protocol before recruiting individuals to the trial. In Sweden, the national ethics committee particularly reviewed the non-information of the control group and found it ethically acceptable.

INTERVENTIONS:
Procedure: Colonoscopy — Once-only colonoscopy screening
  Arms: Colonoscopy screening

SUMMARY:
Colorectal cancer (CRC) is a major burden in western countries. The disease develops from precursor lesions during a long time-interval. Colonoscopy can detect and remove CRC precursor lesions and may thus be effective for CRC prevention. Many national and international health organisations demand evidence from randomised trials to reduce incidence or mortality of the target disease before advocating population-wide cancer screening. However, while colonoscopy screening for the prevention of colorectal cancer is established in the United States and several European countries, no randomised trials exist to quantify the possible benefit of colonoscopy screening. NordICC is a randomised trial investigating the effect of colonoscopy on CRC incidence and mortality.

NordICC is a multicentre, randomised trial in Nordic countries, the Netherlands and Poland. A minimum of 66 000 individuals, age 55-64 years, are drawn randomly from the population registries in the participating countries. 22 000 are invited for once-only colonoscopy (2:1 randomisation). Expected work-load with 50% compliance will be 11,000 colonoscopies. At the screening examination, all detected lesions are biopsied and removed whenever possible. The remaining 44 000 individuals (control group) are not offered any screening examination (care as usual).The primary study aims are CRC incidence and CRC mortality after 15 years of follow-up, with an interim analysis after 10 years of follow-up. In an intention-to-treat approach, a risk reduction of CRC mortality of 25% in the colonoscopy screening group compared to the control group is expected after 10 years follow-up, estimating 50% compliance in the screening group.

ELIGIBILITY:
Inclusion Criteria:

* This study is a population-based randomised controlled trial, with randomisation of individuals age 55-64 years living in the screening areas directly from the Population Registries to either screening group or control group. Eligible persons with the same home address will be randomised to the same group (household randomisation).

Exclusion Criteria:

* Individuals with previous colorectal surgery (resections, enterostomies)
* Individuals in need of long-lasting attention and nursing services (somatic or psychosocial, mental retardation).
* On-going cytotoxic treatment or radiotherapy for malignant disease
* Severe chronic (longer than trial duration) cardiac (NYHA III-IV)or lung disease
* Lifelong anticoagulant therapy with Warfarin
* A coronary event requiring hospitalization during the last 3 months
* A cerebrovascular event during the last 3 months
* Resident abroad
* Return of unopened letter of invitation and/or reminder (address unknown)
* Message from neighbour/family/post office on death of screenee (not updated in Population Registry)

Ages: 55 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95000 (Actual)
Dates: Start 2009-05; Primary Completion 2026-06 (Estimated); Study Completion 2036-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of the screening group vs. the control group in an intention-to-treat model after 15 years of follow-up with regard to CRC mortality and CRC incidence | 15 years after screening (interim analysis after 10 years)

SECONDARY OUTCOMES:
CRC mortality and CRC incidence of screening attendees compared to the control group and non-attendees | 15 years after screening (interim analysis after 10 years)
Mortality from all causes | 15 years after screening (interim analysis after 10 years)

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Olov Adami, MD PhD, Study Director — Harvard School of Public Health, Boston, USA; Michael Bretthauer, MD PhD, Principal Investigator — Oslo University Hospital; Michal Filip Kaminski, MD PhD, Principal Investigator — Marie Cure Sklodowska Cancer Center
Locations (7):
- United States (2):
  - Harvard School of Public Health, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
- Landspitali University Hospital, Reykjavik, Iceland
- Erasmus University Medical Center, Rotterdam, Netherlands
- Oslo University Hospital, Oslo, Norway
- Maria Sklodowska-Curie Memorial Cancer Centre, Warsaw, Poland
- Karolinska Institute, Stockholm, Sweden

REFERENCES:
- [Derived] Bretthauer M, Loberg M, Wieszczy P, Kalager M, Emilsson L, Garborg K, Rupinski M, Dekker E, Spaander M, Bugajski M, Holme O, Zauber AG, Pilonis ND, Mroz A, Kuipers EJ, Shi J, Hernan MA, Adami HO, Regula J, Hoff G, Kaminski MF; NordICC Study Group. Effect of Colonoscopy Screening on Risks of Colorectal Cancer and Related Death. N Engl J Med. 2022 Oct 27;387(17):1547-1556. doi: 10.1056/NEJMoa2208375. Epub 2022 Oct 9. PMID 36214590
- [Derived] Shaukat A, Kahi CJ, Burke CA, Rabeneck L, Sauer BG, Rex DK. ACG Clinical Guidelines: Colorectal Cancer Screening 2021. Am J Gastroenterol. 2021 Mar 1;116(3):458-479. doi: 10.14309/ajg.0000000000001122. PMID 33657038
- [Derived] Bretthauer M, Kaminski MF, Loberg M, Zauber AG, Regula J, Kuipers EJ, Hernan MA, McFadden E, Sunde A, Kalager M, Dekker E, Lansdorp-Vogelaar I, Garborg K, Rupinski M, Spaander MC, Bugajski M, Hoie O, Stefansson T, Hoff G, Adami HO; Nordic-European Initiative on Colorectal Cancer (NordICC) Study Group. Population-Based Colonoscopy Screening for Colorectal Cancer: A Randomized Clinical Trial. JAMA Intern Med. 2016 Jul 1;176(7):894-902. doi: 10.1001/jamainternmed.2016.0960. PMID 27214731
- [Derived] Pisera M, Kaminski MF, Kraszewska E, Rupinski M, Regula J. Reinvitation to screening colonoscopy: a randomized-controlled trial of reminding letter and invitation to educational meeting on attendance in nonresponders to initial invitation to screening colonoscopy (REINVITE). Eur J Gastroenterol Hepatol. 2016 May;28(5):538-42. doi: 10.1097/MEG.0000000000000578. PMID 26967693
- [Derived] Kaminski MF, Bretthauer M, Zauber AG, Kuipers EJ, Adami HO, van Ballegooijen M, Regula J, van Leerdam M, Stefansson T, Pahlman L, Dekker E, Hernan MA, Garborg K, Hoff G. The NordICC Study: rationale and design of a randomized trial on colonoscopy screening for colorectal cancer. Endoscopy. 2012 Jul;44(7):695-702. doi: 10.1055/s-0032-1306895. Epub 2012 Jun 21. PMID 22723185